CLINICAL TRIAL: NCT06291909
Title: Small Steps Towards Personalized Dementia Prevention: Implementation and Evaluation of a Personalized, Technology-assisted Physical Behaviour Intervention
Brief Title: Small Steps Towards Improving Activity and Sleep Habits to Decrease the Risk of Dementia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Australia (Other)
Collaborators: Flinders University (Other)
Responsible Party: Principal Investigator, A/Prof Ashleigh Smith, Associate Professor in Healthy Ageing, UniSA Allied Health & Human Performance, University of South Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 205989
Record Dates: First submitted 2024-02-18; First posted 2024-03-04 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Alzheimer Disease
Keywords: physical activity; sleep; sedentary behavior; behavioral intervention; cognition; dementia
MeSH Terms: conditions — Dementia; Alzheimer Disease; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Condensed Program Group (Placebo Comparator): Identification of optimal time use with comparison to current time use. No research staff supported goal setting, provision of lifestyle information resources through website (no other website functionality available).
  Interventions: Behavioral: Comparator Program
- Extended Program Group (Experimental): Identification of optimal time use with comparison to current time use, complete access to the Small Steps digital interface, frequent one-on-one support from research staff, supported goal setting and behaviour change choices.
  Interventions: Behavioral: Small Steps Program

INTERVENTIONS:
Behavioral: Small Steps Program — Participants in the intervention group will be given access to the Small Steps website. Small Steps website provides a visual representation of the participant's current use of time and allows for manipulation to demonstrate how small lifestyle changes may improve sleep and physical activity needs. The personal outcome goals selected by the participant will also feature on participant's dashboard within the Small Steps website as a reminder. Participants will be prompted through the first 12 weeks to add a new behaviour change each week and will receive support phone calls weekly. During the 12-week Maintenance Phase participants will be guided to maintain their new behaviour, with supportive phone calls being progressively reduced from fortnightly to monthly. At the completion of the 12 weeks, investigator support will be withdrawn. Maintenance of the new behaviour without support will then be assessed over 12 additional weeks in the Follow-Up phase.
  Other Names: Extended Program
  Arms: Extended Program Group
Behavioral: Comparator Program — Participants will receive generic health advice only and it will not be individually tailored, nor will they receive weekly support phone calls during the first 12-weeks. Participants will receive no feedback or support in the Maintenance or Follow-Up phases.
  Other Names: Condensed Program
  Arms: Condensed Program Group

SUMMARY:
This is a randomised controlled study aiming to evaluate the implementation of a website ('Small Steps') to support the modification of participants' time-use behaviour to reduce the risk factors for dementia. 'Small Steps' website provides the tools for this with a visual representation of the participant's current use of time and allowing manipulation to demonstrate how small lifestyle changes may improve and meet sleep and physical activity needs. Participants will be assisted to make changes to current behaviours with the aim to reduce the time they spend sitting (sedentary behaviour), increase physical activity, and improve sleep duration and quality.

Participants (aged 65 or older) will be randomly allocated to one of two groups, the 'Extended Program' (intervention) group or the 'Condensed Program' (control) group.

There are 3 phases (Introductory, Maintenance and Follow-Up; each 12-weeks long) to this program and in total the program is 36-weeks long. Participants will use a tailored website to help support them in making progressive changes over the first 12 weeks. They will then try to maintain these behaviour changes for as long as possible. There will be in-person health testing during each phase and information about sleep habits, sleep quality, and motivation will be assessed using online surveys. Physical activity levels and sleep duration will also be assessed.

DETAILED DESCRIPTION:
The investigators have previously co-designed a personalised, technology-assisted physical activity intervention called 'Small Steps', which promotes positive behaviour changes to reduce dementia risk factors. The current study aims to implement and evaluate this intervention. The 'Small Steps' website provides the tools for facilitating changes in time-use behaviours with a visual representation of the participant's current use of time and allowing manipulation to demonstrate how small lifestyle changes may improve and meet sleep and physical activity needs. Rather than considering single time-use components as independent variables, including 24-hour time-use compositions in the same analytical model will allow the inevitable interplay between the individual components to be assessed.

Older adults most at risk of dementia (older population, low physical activity levels, lower socio-economic status areas) will be recruited. Participants will be assessed face-to-face by trained research staff at study Enrolment, and completion of the Introduction, Maintenance and Follow-Up Phases (each phase is 12 weeks long). The trial will involve comprehensive assessments including detailed demographics, anthropometry and time-use assessments.

The intervention will be modelled on our previously successful method of reducing sitting time in older adults and use recommendations of the optimal activity composition generated from a previous study (ACTIVate Study, Smith et al. BMJ Open 2022;12:e047888). Older adults will be able to work with research staff to co-create interventions that are individualised for their own needs based on individual preferences, constraints and lifestyle. It is hypothesised that the Small Steps intervention will be both more effective than generic health advice (control group) and effects will hold over time (to end of the Follow Up Phase).

Hypotheses: In older adults at risk of dementia, a Small Steps intervention compared to generic health advice will be feasible and associated with:

1. increased time spent in physical activity from Enrolment to end of the each phase, compared to generic health advice.
2. improved cognitive functioning assessed by the Addenbrooke's Cognitive Exam.
3. improved sleep quality as assessed by the Pittsburgh Sleep Quality questionnaire and Sleep Hygiene Index.

Aims:

1) Assess the feasibility of a personalised technology assisted behavioural intervention to improve the 24-hour time use of older adults.

2.) Assess whether a personalised 24-hour time-use intervention increases physical activity and improves sleep behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Ambulatory and community dwelling
* Fluent in the English Language (required for cognitive assessments)
* Resident of City of Onkaparinga Council, Marion City Council, City of Port Adelaide and Enfield, City of Playford, City of Salisbury, City of Tea Tree Gully
* Access and competency in using technology (i.e., phone, tablet, computer)
* Not meeting the Australian physical activity guidelines - 150 minutes per week of moderate intensity physical activity (self-report)
* Deemed safe to participate in physical activity (ESSA APSS stage 1) or clearance from health professional

Exclusion Criteria:

* Scores below the mild cognitive impairment (MCI) cut-off (<13/22) on the Montreal Cognitive Assessment-Blind (MoCA-B) or a current diagnosis of dementia
* Self-reported meeting the Australian physical activity guidelines
* Major neurological or psychiatric diagnosis
* Known intellectual disability
* Major physical disability
* Lack of English fluency
* Involved in another intervention trial involving physical activity, brain training, and/or diet
* Have vision problems which may prevent them from reading a computer and/or phone screen

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participant logins onto the "Small Steps" website | 0-36 weeks
  Analysis of the Small Steps website will be performed to provide the number of logins for each on participant with the 'Small Steps' website. A higher the number of logins, indicates greater engagement with the website.
Number of participant check-ins on the "Small Steps" dashboard | 0-36 weeks
  Analysis of the Small Steps website will be performed to provide the number of check-ins for each on participant with the 'Small Steps' website. Participants are asked to check-in weekly at a minimum. A higher the number of logins, indicates greater engagement with the website.
Number of participant behavioural change choices on the "Small Steps" website during the Introduction Phase. The greater number of choices indicates a greater engagement with the intervention and use of the website. | 0-12 weeks
  Analysis of the Small Steps website will be performed to analyse the number of behavioural change choice each participant makes within the 'Small Steps' website. A higher the number of choices, indicates greater engagement with the intervention.
Time participants spent on the "Small Steps" website | 0-36 weeks
  Analysis of the Small Steps website will be performed to analyse the time each participant spends on the 'Small Steps' website. This will be measured in minutes/login and total number of minutes. A greater number of minutes, indicates greater engagement with the intervention.
Duration of each participant behavioural change choice during the Introductory Phase | 0-12 weeks
  The duration of each behavioural change the participants choose to make at each week. The duration will be measured in minutes/day for each new behavioural change choice.
Holden's Simplified System Usability Scale | 12 and 24 weeks
  The intervention feasibility will be measured by Holden's Simplified System Usability Scale questionnaire, participant reported. The Holden's Simplified System Usability Scale is 10-item design, five-item agreement-based Likert scale, from Strongly agree (5) to Strongly disagree (1) with total scores ranging from 10- 50. It allows you to evaluate software, mobile devices, websites and applications. A higher score indicates greater usability.
Health Care Climate Questionnaire | 12 and 24 weeks
  The intervention acceptability will be measured by the Health Care Climate Questionnaire (participant reported). This is a 6 item (shortened version) using a 7-point Likert-type scale, from Not At All True (1) to Very True (7). The total scores will range from 6 - 42 and a higher score indicates greater acceptability. The preamble and wording of each item will be altered, to better align with the Small Steps intervention and the role of the health professional.
Behavioural Automaticity Questionnaire | 0, 12, 24 and 36 weeks
  The intervention acceptability feasibility will be measured by a Behavioural automaticity (Self-Report Behaviour Automaticity Index) questionnaire. Participants rate items (such as "Physical activity is something I do automatically") on a scale ranging from 1 (strongly disagree) to 7 (strongly agree). Participants will complete the measure in relation to four different behaviours; physical activity, sedentary behaviour, and good sleep practices with each of these 4 behaviours ranging in scores from 4-28. A higher score indicates greater automaticity for that behaviour.
Self-efficacy and Intention Questionnaire | 0, 12, 24 and 36 weeks
  The intervention feasibility will be measured by self-efficacy and intention questionnaire (participant reported). Participants self-efficacy for physical activity will be captured through the self-efficacy for exercise scale. Intention to be physically active and perform positive sleep behaviours will each be assessed. Participants will respond on a 7-point Likert scale with options ranging from 1 (Strongly Disagree) to 7 (Strongly Agree). The total scores will range from 7- 14, with a higher score indicating greater feasibility of the intervention.
Perceived Competence Scale | 0, 12, 24 and 36 weeks
  Participants' satisfaction of their psychological needs of competence will be assessed using the Perceived Competence Scale. This is a short 4-item questionnaire assessing participants' perceived competence to exercise. Participants respond to the 4-items using a 7-point Likert type scale, ranging from 1 (not at all true) to 7 (very true). The total scores will range from 4 - 28, with a higher score indicating greater participant confidence and feelings of competence.
Exit interview | 36 weeks
  A single Semi-structured exit interview will elicit rich data on participant experiences, perceived burden, suggestions for improvement and barriers to feasibility.
Daily activity | 0, 12, 24 and 36 weeks
  Continuous recording using a wrist-worn activity monitor (FitBit) with daily time-use derived from a 7-day average. Time spent in sedentary, light, moderate-to-vigorous and vigorous physical activity (min/day).
Sleep quality | 0, 12, 24 and 36 weeks
  Self-reported sleep quality as measured by Pittsburgh Sleep Quality Index (PSQI). The PSQI is 19-item self-report index to assess sleep quality. The questionnaire consists of a combination of Likert type and open-ended questions (later converted to scaled scores using provided guidelines). Scoring provides an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Sleep Hygiene | 0, 12, 24 and 36 weeks
  Self-reported sleep quality as measured by Sleep Hygiene Index (SHI). The SHI is a 13-item self-report index designed from the ICSD to assess the presence of sleep hygiene behaviours. Each of the item is rated on a five-point Likert scale (ranging from 0 [never] to 4 [always]). The total scores ranged from 0 to 52, with higher scores indicating poorer sleep hygiene status.
Sleep quantity | 0, 12, 24 and 36 weeks
  Continuous recording using a wrist-worn activity monitor (FitBit) with daily time-use derived from a 7-day average with sleep time measured in minutes per day.

SECONDARY OUTCOMES:
Addenbrooke's Cognitive Exam III | 0, 12, 24 and 36 weeks
  Scores for Addenbrooke's Cognitive Exam III (ACE-III). This consists of 19 activities which test five cognitive domains: attention (score 0-18), memory (score 0- 26), fluency (score 0-14), language (score 0 - 26) and visuospatial processing (0-16). The total score is 100 with higher scores indicating better cognitive functioning.
Trail Making Test | 0, 12, 24 and 36 weeks
  Score for Trail Making Test. The Trail Making Test (TMT) is a timed neuropsychological test that involves visual scanning and working memory. The TMT is scored by how long it takes to complete the test (seconds). Norms have been established based on age and education and the lower the number of seconds taken the better the cognitive functioning.
Digit Span Test | 0, 12, 24 and 36 weeks
  Score for Digit Span Test. This test measures short-term verbal memory. The total number of lists reported correctly is combined across forward span (FS) and backward span (BS) to produce a total correct score. Outcome measures include the direction of the task (forwards or backwards), the longest sequence successfully reached and passed, and the total number of attempts. The higher the score the better the cognitive functioning.
24-hour time-use patterns | 0, 12 and 36 weeks
  24-hour time use will be captured via self-report using the Multimedia Activity Recall for Children and Adults (MARCA) tool (30). The MARCA will be conducted via telephone call with a trained researcher and requires participants to recall every activity that they engaged in over the past two days from midnight to midnight, in minimum 5-minute increments. The MARCA tool contains over 500 activities linked to an activity compendium, allowing 24-hour time use to be conceptualised in terms of both activity types and activity intensities (through linking each individual activity with its metabolic equivalent per the compendium).
Measures of behavioural change | 0, 12, 24 and 36 weeks
  Participants' motivation to be physically active will be captured using the Treatment Self-Regulation Questionnaire. Participants will respond to 15 questions relating to reasons for beginning or keeping regular disease self-management, such as "Because I personally think it is best for my health" and "Because I would feel guilty or ashamed if I did not manage my own disease" using a 7-point Likert-type scale (1=not true at all, 7=completely true).

CONTACTS AND LOCATIONS:
Overall Officials: Ashleigh Smith, PhD, Principal Investigator — University of South Australia
Locations (1):
- University of South Australia, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mellow ML, Blake HT, Ferguson T, Robins B, Dumuid D, Olds T, Stanford TE, Laver K, Keage H, Coates A, Wade AT, Rogers M, Davis A, Di Venuto L, Tregoweth E, Yandell C, Tainsh B, Smith AE. 'Small Steps' towards improving 24-hour time-use behaviours to decrease the risk of dementia: protocol for a personalised, web-based randomised controlled trial in community-dwelling older adults. BMJ Open. 2025 Nov 4;15(11):e105643. doi: 10.1136/bmjopen-2025-105643. PMID 41193209